CLINICAL TRIAL: NCT01199328
Title: A Phase I, Open, Two-way Crossover, Drug-drug Interaction Study Evaluating the Effect of Esomeprazole on the Pharmacodynamics of Acetylsalicylic Acid After 5 Days of Treatment
Brief Title: Study to Evaluate the Interaction Between Aspirin and Nexium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MDS, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D961FC00011
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers
Keywords: Nexium; aspirin; peptic ulcers; pharmacodynamic (PD); Esomoeprazole
MeSH Terms: conditions — Peptic Ulcer | interventions — Aspirin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Aspirin 81 mg
  Interventions: Drug: Aspirin
- 2 (Active Comparator): Esomeprazole 20mg/aspirin 81mg
  Interventions: Drug: Aspirin; Drug: Esomeprazole

INTERVENTIONS:
Drug: Aspirin — 81mg Tablet oral, once daily
Drug: Esomeprazole — 20 mg Tablet oral, once daily
  Other Names: Nexium
  Arms: 2

SUMMARY:
The purpose of this study is to assess the interaction between aspirin and Nexium in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 75 years with suitable veins for cannulation or repeated vein puncture.
* Healthy female subjects must be of non-childbearing potential (post-menopausal, had a hysterectomy and/or bilateral oophorectomy) or be of childbearing potential and have a negative serum hCG pregnancy test during screening and be using of the following methods of birth control:
* Continuously practice abstinence during screening and throughout the duration of the study
* Clinically accepted contraception as described under item 7 of Section 5.1 and on hormonal contraceptives.
* Have a body mass index (BMI) between 19 and 30 kg/m2
* No clinically significant abnormal findings as judged by the Investigator on enrollment physical exam.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrolment or randomisation in the present study.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study e.g. history of any bleeding disorder, excessive bruising or ongoing or history of liver disease
* History or presence of clinically significant gastrointestinal e.e. GI ulcer, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness within 4 weeks of the first administration of investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of esomeprazole on low-dose aspirin pharmacodynamics by assessing the relative change in the VerifyNow Aspirin test after 5 days of treatment, relative to baseline (Day 1) in healthy human volunteers | Ongoing throughout the study from consent through withdrawal

SECONDARY OUTCOMES:
Evaluate the effect of esomeprazole on low-dose aspirin pharmacodynamics by assessing the relative change in serum thromboxane B2 inhibition from baseline | Ongoing throughout the study from consent through withdrawal
Evaluate safety and tolerability of esomeprazole taken concurrently with low- dose aspirin | Ongoing throughout the study from consent through withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N Morrison, MD, Principal Investigator — Bio-Kinetic Clinical Applications; Tore Lind, Study Director — AstraZeneca; Lynne Durborow, Study Chair — AstraZeneca
Locations (1):
- Research Site, Springfield, Missouri, United States

REFERENCES:
- [Derived] Andersson T, Morrison D, Nagy P, Pisupati J, Schettler J, Warner TD. Evaluation of the pharmacodynamics of acetylsalicylic acid 81 mg with or without esomeprazole 20 mg in healthy volunteers. Am J Cardiovasc Drugs. 2012 Aug 1;12(4):217-24. doi: 10.1007/BF03261830. PMID 22631032